CLINICAL TRIAL: NCT01555593
Title: Effect of Prolonged Decubitus on Bronchial Inflammation in COPD Patients Evaluated by Expired NO Concentration Assessment
Brief Title: Effect of Prolonged Decubitus on Nitric Oxide Concentration in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Pierachille Santus, Head of Pulmonary Rehabilitation Unit, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 630CEC
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: COPD; FeNO; Bronchial inflammation; Small airways; Decubitus
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COPD FEV1<70%pred feNO Cardioline Exp'air (Experimental): COPD subjects with FEV1<70% of predicted value and Forced Expiratory Volume Forced to Forced Vital Capacity ratio (FEV1/FVC) less than 88% (males)or less than 89% (females) of Low Levels of Normality (LLN) entering the respiratory rehabilitation unit will undergo multiflow feNo measure with Cardioline Exp'air by Medi-soft - Sorinnes (B)
  Interventions: Device: Cardioline Exp'air by Medi-soft - Sorinnes (B)

INTERVENTIONS:
Device: Cardioline Exp'air by Medi-soft - Sorinnes (B) — FeNO measurement in four different moments, the first in the evening, the last three in the morning of the day after. These evaluations will be repeated when the patient enters the unit and after 15 days of rehabilitation activity

SUMMARY:
* Bronchial obstruction in Chronic Obstructive Pulmonary Disease (COPD) is caused by inflammation of peripheral airways walls.
* Neutrophils and other inflammatory mediators Interleukin-6 (IL6), Interleukin-8 (IL8), Interleukin-1 alpha (IL-1 alpha),Interleukin-1beta (IL-1 beta), Tumor Necrosis Factor alfa (TNF-alfa), Reactive Oxygen Species (ROS), Leukotriene B4 (LTB4), Nitric Oxyde (NO) are implicated in the inflammation.
* Exhaled NO concentration is usually used to monitor bronchial inflammation
* The relationship between decubitus and small airways behaviour is not well understood.
* Our hypothesis is that cyclic opening and closure of peripheral airways during decubitus can provoke an inflammatory response which can be monitored by exhaled NO.
* Data about these physiopathological aspects is missing in literature.

DETAILED DESCRIPTION:
Bronchial inflammation in COPD represents one of the main causes of not fully reversible obstruction and airflow limitation. The main inflammatory cells involved are represented by the neutrophils, while some inflammatory mediators (IL6, IL8, IL1alpha, IL1beta, TNFalfa, ROS, LTB4, NO) provoke the disruption of the elastic alveolar bonds that support the small airways, thus invalidating their physical and mechanical characteristics. During decubitus, in such patients, the more dependent parts of the lung are subjected to gravity force, which together with chronic inflammation may cause, we suppose, one of the following effects during tidal breathing:

* a total closure of the smaller bronchioli
* a cyclic opening and closure of the small airways thus provoking friction and an inflammatory response of mechanical origin.

The Fraction of Exhaled Nitric Oxyde (FeNO) concentration is largely used in clinical practice as a marker to monitor the lung inflammatory status.

The purpose of the study is to evaluate the possible mechanical origin of the bronchial inflammation in correlation with prolonged supine decubitus, and so use the NO as an index of the small airways impairment in COPD patients.

To do this we will measure the exhaled NO concentration in COPD patients with moderate to severe obstruction, that is a Forced Expiratory Volume less than 70% of predicted value (FEV1<70%pred). The evaluation will be done in four different moments:

1. before the patient goes to sleep while in supine position
2. immediately after the patient wakes up in the morning, still being in supine position.
3. while sitting on the bed after point 2
4. in the morning after one hour of normal patient's activities, in seated position.

Together with NO concentration, also the Respiratory Frequency and Tidal Volume will be registered during each evaluation.

All the subjects will be inpatients accessing a respiratory rehabilitation unit. At the beginning and after 15 days of rehabilitation a functional respiratory assessment will be made (spirometry, plethysmography, Carbon Monoxide (CO) diffusion lung test), together with an arterial blood gas analysis and a 6 minutes walking test (WT6').

An initial and a final assessment of dyspnoea will be made by Borg and Modified Medical Research Council (mMRC) scales. For the study duration all the patients will continue their inhaled therapy as usual (an ultra long acting anticholinergic once daily plus a long acting Beta-2 agonist in combination with an inhaled corticosteroid twice daily)

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* COPD patients with age raging from 50 to 85 years old
* Patients with at least a history of COPD of one year
* COPD patients clinically stable in the last three months
* COPD subjects with FEV1<70% of predicted value
* FEV1/FVC <88% (males) or <89% (females) of LLN
* COPD former or active smokers with at least a smoking history of 20 pack year

Exclusion Criteria:

* Acute Bronchial Exacerbation at recruitment
* Fertile women with age between 18 and 50 years old or with active period
* Pregnancy
* Subjects enrolled in other clinical trials or that have taken part in one of them in the month preceding the enrollment.
* FEV1/FVC more than 70% of predicted value in basal conditions
* FEV1 more than 70% of predicted value in basal conditions
* Known deficit of alpha 1 antitrypsin
* Subjects that underwent a Lung Volume Reduction Surgery (LVRS)
* Subjects with known positivity to Human Immunodeficiency Virus (HIV)
* Misuse of alcool or drugs
* Lack of compliance in performing respiratory tests
* Subjects not capable to follow the study prescriptions because of psychic disorders or language problems.
* Long Term Oxygen Therapy with flows > 6 litres per minute (l/min) at rest

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change of Fraction of Exhaled Nitric Oxide related to patient's change of decubitus before and after a rehabilitation cycle | The exhaled NO concentration will be assessed in two different moments: the day immediately after the hospitalization (t0) and after 15 days (t1) of rehabilitation activity
  NO concentration will be evaluated in four different sessions at t0 and t1: 1) immediately after the patient goes to bed while he is in supine position; 2) when the patient wakes up, when he's still in the bed in supine position; 3) in sitted position after 5 deep inspirations to total lung capacity 4) after one hour of normal morning activity, again in sitted position. The NO measurements will be collected by a portable NO analyzer at the patient's bed.

CONTACTS AND LOCATIONS:
Overall Officials: Pierachille Santus, Md, PhD, Study Director — Università degli Studi di Milano-Pneumologia Riabilitativa-Fondazione Salvatore Maugeri-MILANO
Locations (1):
- : Pneumologia Riabilitativa-Fondazione Maugeri-Istituto Scientifico di Milano- IRCCS, Milan, Milano, Italy